CLINICAL TRIAL: NCT01248351
Title: Reversibility of Dual Antiplatelet Therapy by Platelets.Phase II Study
Brief Title: Reversibility of Dual Antiplatelet Therapy by Platelets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Novo Nordisk A/S (Industry); CSL Behring (Industry)
Responsible Party: Univ. Prof. Dr. Elisabeth Mahla, Medical University of Graz
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAC_2009; 2009-018108-17 (EudraCT Number)
Record Dates: First submitted 2010-11-19; First posted 2010-11-25 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Bleeding
Keywords: aspirin, clopidogrel, pharmacodynamics, platelet transfusion
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- autologous stored platelets (Experimental)
  Interventions: Other: autologous stored platelets; Other: administration of autologous stored platelets; Biological: autologous stored platelets

INTERVENTIONS:
Other: autologous stored platelets — Administration of autologous stored platelets
Other: administration of autologous stored platelets — administration of autologous stored platelets
Biological: autologous stored platelets — transfusion of autologous stored platelets

SUMMARY:
The objective of the study is to test the hypothesis whether or not autologous stored platelets are able to offset the antiplatelet effect of aspirin and clopidogrel as assessed by state-of-the-art platelet function assays.

DETAILED DESCRIPTION:
Dual antiplatelet therapy with aspirin and clopidogrel is a well established strategy to prevent thrombotic complications in patients with high platelet reactivity following plaque rupture in acute coronary syndromes (ACS) or percutaneous coronary interventions. Current practice guidelines for antiplatelet therapy advocate a one to 12 months dual antiplatelet therapy after bare metal stent PCI and a 12 months dual antiplatelet therapy after PCI in patients with ACS and drug eluting stent PCI. Although oral antiplatelet therapy is associated with both, short- as well as long-term clinical efficacy, irreversible platelet inhibition carries a substantial risk of bleeding particularly in patients presenting for surgery. Empiric therapy of bleeding consists of platelet transfusion. However, there are currently no pharmacodynamic studies assessing the effect of stored platelets on in-vitro platelet function tests.

Healthy volunteers will donate platelets, take aspirin and clopidogrel for 3 days (loading dose aspirin 300 mg, clopidogrel 300 mg, maintenance dose aspirin 100 mg, clopidogrel 75 mg) and platelets will be retransfused on the 4th day. Pharmacodynamic measurements of platelet function will be performed at baseline, after drug intake before retransfusion, immediately after retransfusion and 24 hours thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Healthy volunteers, male or female (after exclusion of pregnancy if they are on birth control pill or have a contraceptive coil implanted)
3. Age of consent
4. Weight: 70 kg - 100 kg
5. Platelet count 240 000 to 440 000/µL
6. Hematocrit > 40%
7. readiness to refrain from any activities prone to injury during the study period.

Exclusion criteria:

1. Allergy against aspirin or clopidogrel
2. History of bleeding
3. History of peptic ulcer
4. Intake of aspirin or NSAR during the last ten days before screening
5. Gastrointestinal disease precluding resorption of aspirin and clopidogrel
6. Scheduled surgery
7. Any current medication
8. History of hepatic disease
9. 20µm ADP induced aggregation < 60% at screening
10. CYP2C19 polymorphisms
11. Donation of blood within the preceding 4 weeks
12. Neurotic disease
13. Current smoking
14. Drug addiction
15. Intake of grapefruits during the last 10 days before

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic assessment of platelet function as assessed by 5 and 20 micromolar ADP | 7 days
  pharmacodynamic measurements of platelet function will be assessed at baseline, after 3 days administration of aspirin and clopidogrel (300 mg loading with aspirin and clopidogrel, maintenance with 100 mg aspirin and 75 mg clopidogrel, respectively) after retransfusion of stored platelets and 24 hours thereafter

SECONDARY OUTCOMES:
Pharmacodynamic assessment of platelet function as assessed by 20 mM arachidonic acid | 7 days
  pharmacodynamic measurements of platelet function will be assessed at baseline, after 3 days administration of aspirin and clopidogrel (300 mg loading with aspirin and clopidogrel, maintenance with 100 mg aspirin and 75 mg clopidogrel, respectively) after retransfusion of stored platelets and 24 hours thereafter
Pharmacodynamic assessment of platelet function as assessed by Vasodilator stimulated phosphoprotein (VASP) phosphorylation (platelet reactivity index; PRI) | 7 days
  pharmacodynamic measurements of platelet function will be assessed at baseline, after 3 days administration of aspirin and clopidogrel (300 mg loading with aspirin and clopidogrel, maintenance with 100 mg aspirin and 75 mg clopidogrel, respectively) after retransfusion of stored platelets and 24 hours thereafter
Pharmacodynamic assessment of platelet function as assessed by expression of GP IIb/IIIa receptors and P-selectin (Mean fluorescence intensity %) | 7 days
  pharmacodynamic measurements of platelet function will be assessed at baseline, after 3 days administration of aspirin and clopidogrel (300 mg loading with aspirin and clopidogrel, maintenance with 100 mg aspirin and 75 mg clopidogrel, respectively) after retransfusion of stored platelets and 24 hours thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Mahla Elisabeth, MD, Principal Investigator — Dept. of Anesthesia and Intensive Care Medicine, Medical University of Graz
Locations (1):
- Department of anesthesia and intensive care medicine, Medical Univerity of Graz, Graz, Austria

REFERENCES:
- [Derived] Pruller F, Drexler C, Archan S, Macher S, Raggam RB, Mahla E. Low platelet reactivity is recovered by transfusion of stored platelets: a healthy volunteer in vivo study. J Thromb Haemost. 2011 Aug;9(8):1670-3. doi: 10.1111/j.1538-7836.2011.04392.x. No abstract available. PMID 21649849